CLINICAL TRIAL: NCT04213807
Title: A Randomized, Placebo-controlled, Dose-range Finding Study to Assess the Pharmacokinetic and Pharmacodynamic Parameters, Safety, Tolerability, and Immunogenicity of MAA868 in Patients With Atrial Fibrillation
Brief Title: A Dose-range Finding Study of MAA868 in Patients With Atrial Fibrillation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anthos Therapeutics, Inc. (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ANT-004
Record Dates: First submitted 2019-12-23; First posted 2019-12-30 (Actual); Results first posted 2021-12-07 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; flutter; paroxysmal atrial fibrillation; stroke; cardiac arrhythmia
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Arrhythmias, Cardiac

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MAA868 (Experimental): Subcutaneous injection on Day 1 with two subsequent monthly injections
  Interventions: Biological: MAA868 Cohort 1; Biological: MAA868 Cohort 2; Biological: MAA868 Cohort 3
- Placebo (Placebo Comparator): Subcutaneous injection: Placebo on Day 1 with two subsequent monthly injections
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: MAA868 Cohort 1 — Subcutaneous injection: low dose
  Arms: MAA868
Biological: MAA868 Cohort 2 — Subcutaneous injection: high dose
  Arms: MAA868
Biological: MAA868 Cohort 3 — Subcutaneous injection: Dose to be determined.
  Arms: MAA868
Other: Placebo — Subcutaneous injection: Placebo
  Arms: Placebo

SUMMARY:
This study is a multicenter, randomized, subject and Investigator-blinded, placebo-controlled, parallel-group, multiple ascending dose-ranging study to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) effects of MAA868 in patients with atrial fibrillation (AF) or flutter at low risk of thromboembolic stroke or peripheral embolism.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥ 18 and < 85 years old with paroxysmal atrial fibrillation (PAF) or atrial flutter on 12 lead electrocardiography at Screening Or
* Patients with a history of PAF or atrial flutter, as documented by (telemetry, 12 lead electrocardiography or ambulatory [e.g. Holter] monitor) and not due to a reversible condition (e.g. alcohol binge drinking) can be entered even if they do not have PAF at Screening. There is not time-limit for this.
* Patients with a Congestive heart failure, Hypertension, Age ( > 65 = 1 point, > 75 = 2 points), Diabetes, previous Stroke/transient ischemic attack (2 points) (CHA2DS2-VASc) risk score (tool as a predictor for estimating the risk of stroke in patients with atrial fibrillation (AF); Lip et al 2010) of 0-1 for men and 1-2 for women and in whom, in the investigator's judgment, the use of an anticoagulant for stroke prevention is not indicated

Exclusion Criteria:

* History of stroke, transient ischemic attack or systemic embolism
* History of major bleeding during treatment with an anticoagulant or antiplatelet therapy. (Patients who have had major bleeding on anticoagulants or antiplatelet therapy more than a year ago can be enrolled only if the bleeding was due to a reversible cause, e.g. gastro-duodenal ulcer that was successfully treated.)
* History of traumatic or non-traumatic intracranial, intraspinal or intraocular bleeding
* Known bleeding diathesis or any known active bleeding site at screening or baseline
* Family history of bleeding disorder
* Known active GI lesions predisposing to bleeding events
* Myocardial infarction, unstable angina pectoris or coronary artery bypass graft (CABG) surgery within 12 months prior to the Screening period
* Known clinically significant valvular heart disease including moderate or severe mitral stenosis (valve area <1.5 cm2)
* Patients with a prosthetic heart valve

Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2020-12-29 (Actual); Study Completion 2021-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman E Lepor, MD FACC FAHA FSCAI, Principal Investigator — Westside Medical Associates of Los Angeles
Locations (6):
- United States (6):
  - Anthos Investigative Site, Beverly Hills, California
  - Anthos Investigative Site, Wichita, Kansas
  - Anthos Investigative Site, Alexandria, Louisiana
  - Anthos Investigative Site, Lansing, Michigan
  - Anthos Investigative Site, Wynnewood, Pennsylvania
  - Anthos Investigative Site, McKinney, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: No subjects were enrolled in the optional Cohort 3.
Pre-assignment Details: 28 participants were screened. 5 participants did not meet inclusion/exclusion criteria; 5 eligible participants failed randomization.
Groups:
- Placebo: Subcutaneous injection of placebo on Day 1, Day 31, and Day 61
- MAA868 120 mg: Subcutaneous injection of 120 mg MAA868 on Day 1, Day 31, and Day 61
- MAA868 180 mg: Subcutaneous injection of 180 mg MAA868 on Day 1, Day 31, and Day 61
Period: Overall Study
Arm/Group | Placebo | MAA868 120 mg | MAA868 180 mg
Started | 5 | 6 | 7
Completed | 5 | 6 | 6
Not Completed | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | MAA868 120 mg | MAA868 180 mg | Total
Number analyzed (Participants) | 5 | 6 | 7 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (18.79) | 53.8 (9.24) | 58.1 (8.34) | 55.1 (11.81)
Age, Customized [Number; unit: years]
  18 to 20 | 1 | 0 | 0 | 1
  21 to 30 | 0 | 0 | 0 | 0
  31 to 40 | 0 | 1 | 0 | 1
  41 to 50 | 0 | 0 | 1 | 1
  51 to 60 | 2 | 4 | 4 | 10
  61 to 70 | 2 | 1 | 2 | 5
  71 to 80 | 0 | 0 | 0 | 0
  81 to 85 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 2 | 5
  Male | 5 | 3 | 5 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 6 | 7 | 18
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 2
  White | 5 | 6 | 5 | 16
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: centimeters] | 182.01 (5.573) | 174.60 (11.311) | 175.74 (8.337) | 177.10 (8.918)
Weight [Mean (Standard Deviation); unit: kg] | 99.352 (13.1715) | 91.667 (7.1102) | 94.933 (23.2745) | 95.072 (16.0115)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 30.022 (4.1647) | 30.392 (4.7558) | 30.887 (8.6754) | 30.482 (6.1179)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Achieved More Than or Equal to 50%, 80%, and 90% Factor XI Inhibition at Trough After the Third Dose (Day 91) at Different Dose Levels of MAA868
Description: Number of participants achieving more than or equal to 50%, 80%, and 90% inhibition of factor XI (less than 50%, 20%, or 10% free factor XI) at trough after the third dose on Day 91 at different dose levels of MAA868
Time Frame: Day 91
Population: Pharmacokinetic/Pharmacodynamic Set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MAA868 120 mg | MAA868 180 mg
Number analyzed (Participants) | 5 | 6 | 7
Participants
  More than or equal to 50% inhibition of factor XI | 0 | 2 | 4
  More than or equal to 80% inhibition of factor XI | 0 | 0 | 1
  More than or equal to 90% inhibition of factor XI | 0 | 0 | 0

2. Secondary Outcome: Number of Participants Achieving More Than or Equal to 50%, 80%, and 90% Factor XI Inhibition at Trough After First (Day 31) and Second Doses (Day 61) at Different Dose Levels of MAA868
Description: Number of participants achieving more than or equal to 50%, 80%, and 90% inhibition of factor XI (less than 50%, 20%, or 10% free factor XI) at trough on Day 31 (after first dose) and Day 61 (after second dose) at different dose levels of MAA868
Time Frame: Day 31 and Day 61
Population: Pharmacokinetic/Pharmacodynamic Set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MAA868 120 mg | MAA868 180 mg
Number analyzed (Participants) | 5 | 6 | 7
Participants
  More than or equal to 50% factor XI inhibition : Day 31 | 0 | 1 | 5
  More than or equal to 50% factor XI inhibition : Day 61 | 0 | 2 | 5
  More than or equal to 80% factor XI inhibition : Day 31 | 0 | 1 | 3
  More than or equal to 80% factor XI inhibition : Day 61 | 0 | 0 | 1
  More than or equal to 90% factor XI inhibition : Day 31 | 0 | 0 | 0
  More than or equal to 90% factor XI inhibition : Day 61 | 0 | 0 | 0

3. Secondary Outcome: Overall Number of Participants Who Experienced Adverse Events, Including Serious Adverse Events, During the Treatment Period and Through End of Study
Description: Overall number of participants who experienced adverse events following multiple subcutaneous administration of MAA868 compared to placebo in participants with atrial fibrillation or atrial flutter
Time Frame: Day 1 through end of study, up to 170 days
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MAA868 120 mg | MAA868 180 mg
Number analyzed (Participants) | 5 | 6 | 7
Participants | 4 | 5 | 3

4. Secondary Outcome: Incidence of Major Bleeding Events, Clinically Relevant Non-major Bleeding Events and Total Bleeding With MAA868 Relative to Placebo
Description: Occurrence of confirmed major bleeding events, clinically relevant non-major bleeding events and total bleeding events during the treatment period
Time Frame: Day 1 through end of study, up to 170 days
Population: Safety Set
Measure: Number; unit: incidence of events
Arm/Group | Placebo | MAA868 120 mg | MAA868 180 mg
Number analyzed (Participants) | 5 | 6 | 7
incidence of events
  Major bleeding events | 0 | 0 | 0
  Clinically relevant non-major bleeding events | 0 | 0 | 0
  Nuisance (not clinically relevant) bleeding events | 2 | 1 | 1
  No bleeding events | 0 | 1 | 0

5. Secondary Outcome: Immunogenicity of MAA868
Description: Number of participants with anti-drug (MAA868) antibodies for all participants who received MAA868 120 mg or MAA868 180 mg.
  "Non-evaluable observation" refers to participants who had no sample collected (due to no visit or remote visit) or for whom the sample was not frozen.
Time Frame: Days 1, 31, 61, 71, 91, 121 and 170
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | MAA868 120 mg | MAA868 180 mg
Number analyzed (Participants) | 6 | 7
Participants
  Baseline: Negative | 6 | 7
  Baseline: Positive | 0 | 0
  Baseline: Non-evaluable observation | 0 | 0
  Day 1: Negative | 6 | 7
  Day 1: Positive | 0 | 0
  Day 1: Non-evaluable observation | 0 | 0
  Day 31: Negative | 6 | 7
  Day 31: Positive | 0 | 0
  Day 31: Non-evaluable observation | 0 | 0
  Day 61: Negative | 3 | 6
  Day 61: Positive | 0 | 0
  Day 61: Non-evaluable observation | 3 | 1
  Day 71: Negative | 4 | 6
  Day 71: Positive | 0 | 0
  Day 71: Non-evaluable observation | 2 | 1
  Day 91: Negative | 5 | 5
  Day 91: Positive | 0 | 0
  Day 91: Non-evaluable observation | 1 | 2
  Day 121: Negative | 5 | 5
  Day 121: Positive | 0 | 0
  Day 121: Non-evaluable observation | 1 | 2
  Day 170: Negative | 6 | 7
  Day 170: Positive | 0 | 0
  Day 170: Non-evaluable observation | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event information was collected at every study visit from providing written informed consent for participation in the study (on Days -28 to -3) until Day 170 (the end of study visit).
Description: The occurrence of adverse events was to be sought by non-directive questioning of the participants at each visit by the site staff during the study (e.g., "How are you feeling today?" or "How have you been feeling since your last visit") to elicit adverse event information from the participant. Adverse events might have been detected when they were volunteered by the participants during or between visits or through physical examination finding, laboratory test finding, or other assessments.
Arm/Group | Placebo | MAA868 120 mg | MAA868 180 mg
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 4/5 | 5/6 | 3/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=5) | MAA868 120 mg (N=6) | MAA868 180 mg (N=7)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Coagulation test abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Eosinophil count increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator agrees that no submission for publication or public disclosure by the Investigator will be made until after publication of the results of the Multicenter Trial, except as set forth in the clinical trial agreement. If, however, there is no multicenter publication within eighteen (18) months after completion or termination of the Study, Investigator may publish or publicly present the Study Data in accordance with the clinical trial agreement.

DOCUMENTS (2):
  • Study Protocol (2020-05-10): https://cdn.clinicaltrials.gov/large-docs/07/NCT04213807/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-18): https://cdn.clinicaltrials.gov/large-docs/07/NCT04213807/SAP_001.pdf